CLINICAL TRIAL: NCT03474250
Title: Trans-catheter Aortic Valve Replacement and Renal Infarction Among Patients With Severe Aortic Stenosis
Brief Title: Trans-aortic Valve Replacement and Renal Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Amit Segev, Proffesor, Sheba Medical Center
Other Study IDs: 4887-18
Record Dates: First submitted 2018-02-22; First posted 2018-03-22 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Renal Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance test for kidney — Magnetic Resonance test for kidney

SUMMARY:
Kidney Magnetic Resonance assessment before and after undergoing transcatheter aortic valve replacement

DETAILED DESCRIPTION:
Each patient will undergo Magnetic Resonance assessment of the kidneys before the TAVR. on the third to 7th day after the ATVR, a second MRI to the kidneys will be performed. we will assess the changes and new lesions between both MRI tests and will perform a qualitative and quantitative measurement.

ELIGIBILITY:
Inclusion Criteria:

* Severe symptomatic aortic stenosis
* Patient is able to lay down supine for 20 min (the time needed to perform the MRI) without any difficulties.

Exclusion Criteria:

* Patient is on chronic renal replacement therapy (Dialysis)
* Documented Thrombus in the left ventricle or left atria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that will be undergoing trans-cather aortic valve replacement for severe symptomatic aortic stenosis
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
New Renal Infarction | one year
  New low signal intensity lesions on diffusion weighted images on MRI.

SECONDARY OUTCOMES:
Hematuria | one year
  New hematuria on urine test.
Elevation in Blood Pressure | one year
  Delta of more than 5%
Elevation in Plasma Renin Activity | one year
  Delta of more than 5%
Elevation in Aldosteron level | one year
  Delta of more than 5%

CONTACTS AND LOCATIONS:
Overall Officials: Arwa Younis, Doctor, Principal Investigator — Tel Aviv University
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided